CLINICAL TRIAL: NCT07205497
Title: Iparomlimab and Tuvonralimab (QL1706) Combined With Neoadjuvant Chemotherapy Followed by Type I Hysterectomy for Locally Advanced Cervical Cancer（QNACTH）: A Prospective, Single-Arm, Multicenter, Phase 2 Trial
Brief Title: QL1706 Plus Neoadjuvant Chemotherapy Followed by Type I Hysterectomy for Locally Advanced Cervical Cancer
Acronym: QNACTH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-206-01
Record Dates: First submitted 2025-04-01; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-03

CONDITIONS: Neoadjuvant Immunotherapy; Locally Advanced Cervical Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eparbrutinib (QL1706) + cisplatin and albumin-bound paclitaxel (Experimental): Participants will take eparbrutinib (QL1706) alongside cisplatin and albumin-bound paclitaxel (TC) every three weeks for three cycles. If the lesion was reduced to less than or equal to 2cm, conectomy was performed; if the pathological results indicated no high-risk factors, total hysterectomy was performed, and QL1706+TC was treated after surgery. If the lesion is larger than 2cm, a type III hysterectomy is performed and adjuvant treatment is determined according to sedlis criteria after surgery.
  Interventions: Drug: QL1706+TC

INTERVENTIONS:
Drug: QL1706+TC — Participants will take eparbrutinib (QL1706) alongside cisplatin and albumin-bound paclitaxel (TC) every three weeks for three cycles. If the lesion was reduced to less than or equal to 2cm, conectomy was performed; if the pathological results indicated no high-risk factors, total hysterectomy was performed, and QL1706+TC was treated after surgery. If the lesion is larger than 2cm, a type III hysterectomy is performed and adjuvant treatment is determined according to sedlis criteria after surgery.

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of the combination therapy of Eparbrutinib (QL1706) with neoadjuvant chemotherapy followed by Type I hysterectomy in treating locally advanced cervical cancer. Additionally, it will assess the safety profile of this treatment regimen. The main questions it aims to answer are:

1. Does the combination of Eparbrutinib (QL1706) with neoadjuvant chemotherapy lead to a higher rate of complete pathological response (pCR) compared to chemotherapy alone?
2. What are the medical complications and side effects experienced by participants during the treatment with Eparbrutinib (QL1706)?

Researchers will compare the outcomes of patients receiving Eparbrutinib (QL1706) combined with neoadjuvant chemotherapy to those receiving standard treatment to evaluate the effectiveness in treating locally advanced cervical cancer.

Participants will:

1. Take Eparbrutinib (QL1706) alongside cisplatin and albumin-bound paclitaxel every three weeks for three cycles.
2. If the lesion was reduced to less than or equal to 2cm, conectomy was performed; if the pathological results indicated no high-risk factors, total hysterectomy was performed, and QL1706+TC was treated after surgery. If the lesion is larger than 2cm, a type III hysterectomy is performed and adjuvant treatment is determined according to sedlis criteria after surgery.
3. Visit the clinic regularly for checkups, tests, and assessments throughout the treatment period.
4. Keep a diary of their symptoms, side effects, and any changes in their health status.

This study is designed to provide insights into the potential benefits of adding Eparbrutinib (QL1706) to the standard neoadjuvant chemotherapy regimen for locally advanced cervical cancer, which may lead to improved treatment outcomes and survival rates for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with untreated cervical cancer at stages IB3, IIA2, and resectable IIIC1r (according to the FIGO standards of 2018; determined by two senior physicians or above through gynecological examination and imaging studies);
2. At baseline, there is at least one measurable tumor lesion according to the RECIST 1.1 criteria, with the size of the lesion primarily determined by magnetic resonance imaging;
3. Pathologically confirmed cervical cancer, including squamous cell carcinoma (all grades), common type adenocarcinoma (Silva classification types A or B, or differentiated grades G1 or G2), and adenosquamous carcinoma (differentiated grades G1 or G2);
4. Patients must be aged between 18 and 70 years inclusive;
5. ECOG performance status score of 0 or 1;
6. Laboratory tests: White blood cell count (WBC) ≥ 3.5 × 10^9/L, neutrophil count (NEU) ≥ 1.5 × 10^9/L, platelet count (PLT) ≥ 100 × 10^9/L, serum bilirubin ≤ 1.5 times the upper limit of normal, transaminases ≤ 1.5 times the upper limit of normal, blood urea nitrogen (BUN) and creatinine (Cr) within normal limits;
7. Capable of follow-up and good compliance;
8. Able to sign an informed consent form, including adherence to the requirements and restrictions listed in the informed consent and this protocol.

Exclusion Criteria:

1. Participants with active, known, or suspected autoimmune diseases, or a history of autoimmune diseases, except for the following conditions: vitiligo, alopecia, Graves' disease, psoriasis, or eczema that does not require systemic treatment within the last 2 years, asymptomatic hypothyroidism or requiring only a stable dose of hormone replacement therapy (due to autoimmune thyroiditis), type 1 diabetes requiring only a stable dose of insulin replacement therapy, asthma that has completely resolved in childhood and does not require intervention in adulthood, or diseases that do not relapse without external triggers;
2. Previously treated with immune checkpoint inhibitors, including but not limited to other anti-PD-1, anti-PD-L1 antibodies, CTLA-4 antibodies, or any treatments targeting immune co-stimulatory factors (such as antibodies targeting ICOS, CD40, CD137, GITR, OX40, etc.) or other mechanisms of tumor immunotherapy;
3. Known allergic reactions to any components and/or excipients of the investigational medication;
4. Received immunosuppressive drugs or systemic corticosteroids for immunosuppression within 2 weeks prior to the study medication (more than 10mg/day of prednisone or other equivalent drugs), with the exception of local, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids;
5. Received traditional Chinese medicine with antitumor effects or drugs with immunomodulatory effects (such as thymic peptides, interferons, interleukin-2) within 2 weeks prior to the study;
6. Active systemic infections requiring systemic treatment;
7. Experienced severe infections within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia;
8. Untreated chronic hepatitis B patients, or hepatitis B virus (HBV) carriers with HBV DNA greater than 1000 IU/mL, or patients with active hepatitis C. Non-active HBsAg carriers, treated and stable hepatitis B patients (HBV DNA < 1000 IU/mL), and cured hepatitis C patients are eligible. Subjects with positive HCV antibodies are only eligible if HCV RNA testing is negative;
9. Known active pulmonary tuberculosis (TB), suspected active TB patients should undergo chest X-ray and sputum tests, combined with clinical symptoms and signs to rule out;
10. Immunodeficiency or human immunodeficiency virus (HIV antibody positive);
11. Participants with active inflammatory bowel disease or a history of such diseases (such as Crohn's disease, ulcerative colitis, or chronic diarrhea). Participants who cannot swallow or have malabsorption syndrome, uncontrolled nausea, vomiting, diarrhea, or other gastrointestinal diseases that severely affect drug intake and absorption;
12. Known interstitial lung disease, symptomatic or likely to hinder the detection or treatment of immune-related pneumonia;
13. Received live vaccines or attenuated vaccines within 4 weeks prior to the first trial dose, with the exception of inactivated seasonal influenza vaccines;
14. Patients who have undergone allogeneic bone marrow transplantation or solid organ transplantation;
15. History of primary malignant tumors within the last 5 years;
16. Participants who have undergone major surgery (such as laparotomy, thoracotomy, organ resection, etc.) and severe trauma within 28 days prior to the first dose, with the exception of implantable infusion devices;
17. History of gastrointestinal perforation, gastrointestinal fistula, or female genital fistula;
18. Uncontrolled other comorbidities, symptoms, or medical history, including: ① Those with one of the following cardiovascular or cerebrovascular diseases or risk factors: myocardial infarction, unstable angina, pulmonary embolism, acute/persistent myocardial ischemia, cerebrovascular accident, transient ischemic attack, or other clinically significant/requiring medication intervention arterial venous thrombosis, embolism, or cerebral ischemic events; symptoms of congestive heart failure within 6 months (New York Heart Association (NYHA) class III or above); ② History of clinically significant bleeding symptoms or obvious bleeding features within 1 month prior to the first dose, such as gastrointestinal bleeding, peptic ulcer bleeding, or vasculitis; ③ Clinical manifestations of active hemoptysis, active diverticulitis, abdominal abscess, and gastrointestinal obstruction; ④ Those with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; ⑤ History of liver or kidney abnormalities or surgery;
19. Pregnant or nursing women; women of childbearing age who refuse to accept contraceptive measures during neoadjuvant immunotherapy;
20. Simultaneously participating in other interventional clinical trials, participation in observational and non-interventional clinical trials is allowed;
21. Any condition deemed by the investigator to pose a risk when receiving the study medication, or that would interfere with the safety evaluation of the study medication or the interpretation of the study results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Within one month after the third cycle of therapy ended (each cycle is 21 days)
  Pathological complete response rate

SECONDARY OUTCOMES:
Rate of conversion to low-risk cervical cancer after treatment | Within one month after the third cycle of therapy ended (each cycle is 21 days)
  Rate of conversion to low-risk cervical cancer after treatment
ORR | Within one month after the third cycle of therapy ended (each cycle is 21 days)
  Objective remission rate
OS | 5 years after the end of the last treatment
  Overall survival
EFS | 5 years after the end of the last treatment
  Event free survival
PFS | 5 years after the end of the last treatment
  Progression free survival
AE | During (3 months) and after the treatment (up to 1 year)
  Adverse event
SAE | During (3 months) and after the treatment (up to 1 year)
  Serious adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- The Sun Yat-sen Memorial Hospital of the Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: When the trial is over and the relevant data has been published.
Access Criteria: With the consent of the corresponding authors.

REFERENCES:
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Park JY, Kim DY, Kim JH, Kim YM, Kim YT, Nam JH. Outcomes after radical hysterectomy according to tumor size divided by 2-cm interval in patients with early cervical cancer. Ann Oncol. 2011 Jan;22(1):59-67. doi: 10.1093/annonc/mdq321. Epub 2010 Jul 1. PMID 20595451
- [Background] GRAY LA, BARNES ML, LEE JJ. Carcinoma-in-situ and dysplasia of the cervix. Ann Surg. 1960 Jun;151(6):951-60. doi: 10.1097/00000658-196006000-00019. No abstract available. PMID 13829114
- [Background] Covens A, Rosen B, Murphy J, Laframboise S, DePetrillo AD, Lickrish G, Colgan T, Chapman W, Shaw P. Changes in the demographics and perioperative care of stage IA(2)/IB(1) cervical cancer over the past 16 years. Gynecol Oncol. 2001 May;81(2):133-7. doi: 10.1006/gyno.2001.6158. PMID 11330939
- [Background] Jing H, Xiuhong W, Ying Y, Zhenrong L, Xiyun C, Deping L, Changmei S, Qi W, Tao P, Yiyun P. Neoadjuvant chemotherapy combined with radical surgery for stage IB2/IIA2 cervical squamous cell carcinoma: a prospective, randomized controlled study of 35 patients. World J Surg Oncol. 2021 Jul 12;19(1):209. doi: 10.1186/s12957-021-02318-y. PMID 34253208
- [Background] Gadducci A, Cosio S. Neoadjuvant Chemotherapy in Locally Advanced Cervical Cancer: Review of the Literature and Perspectives of Clinical Research. Anticancer Res. 2020 Sep;40(9):4819-4828. doi: 10.21873/anticanres.14485. PMID 32878770
- [Background] Gupta S, Maheshwari A, Parab P, Mahantshetty U, Hawaldar R, Sastri Chopra S, Kerkar R, Engineer R, Tongaonkar H, Ghosh J, Gulia S, Kumar N, Shylasree TS, Gawade R, Kembhavi Y, Gaikar M, Menon S, Thakur M, Shrivastava S, Badwe R. Neoadjuvant Chemotherapy Followed by Radical Surgery Versus Concomitant Chemotherapy and Radiotherapy in Patients With Stage IB2, IIA, or IIB Squamous Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Jun 1;36(16):1548-1555. doi: 10.1200/JCO.2017.75.9985. Epub 2018 Feb 12. PMID 29432076
- [Background] Nagano H. Comment on 'Phase III randomised controlled trial of neoadjuvant chemotherapy plus radical surgery vs radical surgery alone for stages IB2, IIA2, and IIB cervical cancer: a Japan Clinical Oncology Group trial (JCOG 0102)'. Br J Cancer. 2013 Oct 29;109(9):2505. doi: 10.1038/bjc.2013.581. Epub 2013 Sep 24. No abstract available. PMID 24064973